CLINICAL TRIAL: NCT03956043
Title: Diagnostic Accuracy of Clinical and Paraclinical Tools in Sepsis
Brief Title: Diagnostic Accuracy in Sepsis
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Aleksander Rygh Holten, Principal Investigator, Oslo University Hospital
Other Study IDs: Sepsis-OUH
Record Dates: First submitted 2019-05-15; First posted 2019-05-20 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Sepsis Syndrome
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with suspected sepsis in Emergency Department: Patients with suspected sepsis treated by the sepsis emergency team or the medical emergency team in the Emergency Department of Oslo University Hospital Oslo are included prospectively.

SUMMARY:
The sepsis syndrome has recently been more stringently defined as "a life-threatening organ dysfunction caused by a dysregulated host response to infection". Clinical and paraclinical tools are investigated for their ability to adequately recognize sepsis early.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old with suspected sepsis in the Emergency Department of Oslo University Hospital Oslo

Exclusion Criteria:

* Non

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oslo University Hospital is a secondary and tertiary Hospital in Norway's largest city Oslo. The Emergency Department treats about 30 000 patient per year, including approximately 500 with suspected sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 1989 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy in sepsis | within 90 days after inclusion
  Sensitivity, specificity, predictive values, AUC of clinical criteria of sepsis in the Emergency department, compared to post hoc assesment
Prognostic accuracy in sepsis | 90 days after inclusion
  Sensitivity, specificity, predictive values, AUC of clinical criteria of sepsis in the Emergency department, compared to in hospital, 30 and 90 days mortality

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander R Holten, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christensen EE, Binde C, Leegaard M, Tonby K, Dyrhol-Riise AM, Kvale D, Amundsen EK, Holten AR. DIAGNOSTIC ACCURACY AND ADDED VALUE OF INFECTION BIOMARKERS IN PATIENTS WITH POSSIBLE SEPSIS IN THE EMERGENCY DEPARTMENT. Shock. 2022 Oct 1;58(4):251-259. doi: 10.1097/SHK.0000000000001981. Epub 2022 Sep 6. PMID 36130401